CLINICAL TRIAL: NCT01330615
Title: A Double-Blind, Randomized, Placebo-Controlled Trial of Eutectic Lidocaine/Prilocaine Cream 5% (EMLA) for Analgesia Prior to Cryotherapy of Verrucae Plantaris in Adults
Brief Title: Efficacy Trial of Eutectic Lidocaine/Prilocaine Cream 5% (EMLA) for Analgesia Prior to Cryotherapy of Verrucae Plantaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Aw Chen Wee, National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: DSRB-E/09/612
Record Dates: First submitted 2010-05-13; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Plantar Warts
Keywords: EMLA; plantar warts; cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryotherapy with EMLA (Active Comparator): EMLA applied before cryotherapy
  Interventions: Drug: EMLA
- Cryotherapy with placebo analgesia (Placebo Comparator): Placebo cream applied instead of EMLA
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EMLA — The cream is applied as a thick layer to the wart and to the surrounding 1 to 2 mm and left on for 60 minutes under occlusion of Tegaderm dressing. The cream is then removed, and liquid cryotherapy applied using cryospray.
  Other Names: Eutectic lidocaine/prilocaine cream 5%
  Arms: Cryotherapy with EMLA
Drug: Placebo — The cream is applied as a thick layer to the wart and to the surrounding 1 to 2 mm and left on for 60 minutes under occlusion of Tegaderm dressing. The cream is then removed, and liquid cryotherapy applied using cryospray.
  Other Names: Dummy treatment, dummy cream
  Arms: Cryotherapy with placebo analgesia

SUMMARY:
Aims:

The investigators main purpose is to assess the efficacy of analgesia provide by topical lidocaine/prilocaine cream 5% (EMLA)® to pared plantar warts prior to application of liquid nitrogen cryotherapy in adults.

DETAILED DESCRIPTION:
Methodology:

The study is a single-centre, double-blind, randomized, placebo-controlled, parallel-group trial with one visit. The investigators planned to include at least 64 patients in 4 months. Adult patients (at least 21 years old) diagnosed with plantar warts are potential subjects for the study.

Once a potential subject is identified, the field investigator will assess him/her for eligibility to enter the study. Then, the potential subject will be provided with full and adequate verbal and written information about the nature, purpose, possible risks and benefits of the study. If the subject agrees to enroll into the study, a signed informed consent will be obtained from him/her.

All patients are randomly assigned by computer-generated randomization sequence to receive either eutectic lidocaine/prilocaine cream (EMLA)® 5% or placebo 60 mins prior to application of cryotherapy. The plantar warts are pared with shape blade before applying EMLA®or placebo cream. Based on the randomization, an designated dermatology laboratory technician will apply either the EMLA® cream 5% or placebo cream to the wart lesions. The cream is applied as a thick layer to the wart and to the surrounding 1 to 2 mm and left on for 60 minutes under occlusion of Tegaderm dressing. The cream is then removed, and liquid cryotherapy applied using cryospray. The lesions are treated with double freeze-thaw cycle. The end point of each freeze is a complete ice-ball covering the lesion with 1-2mm peripheral extension. The study involved only one treatment with either placebo or EMLA® cream 5% followed by cryotherapy as described. No other analgesic other than the EMLA® cream 5% or placebo is allowed at least 2 hours prior to or during cryotherapy.

A 100 mm visual analogue pain scale (VAS) is used to denote pain severity ranging from "no pain" (0 mm) to the "worst possible pain" (100 mm). The patient will choose a distance from the "no pain" anchor closest to the pain experienced during cryotherapy for wart removal. Pain is evaluated in each participant using a self-administered VAS immediately after cryotherapy treatment.

Potential Benefits:

The potential benefits are:

1. The patients may experience less pain during application cryotherapy.
2. The application of local anesthetic cream may possibly increase the effectiveness of cryotherapy.

Potential Risks:

EMLA cream® is known to be relatively safe with minimal side effects. The commonest side effect would be local irritation to the skin e.g. redness, itchiness which is reversible after removal of the cream. Very rarely (<1000), severe allergic reaction can occur with application of EMLA cream® (AstraZeneca information brochure).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (at least 21 years old) with plantar warts
2. They must agree for liquid nitrogen cryotherapy for treatment of the plantar warts
3. The patients have to be capable of assessing pain using a visual analogue pain scale (VAS)

Exclusion Criteria:

1. Patients who had previously used EMLA cream® prior to cryotherapy of warts
2. Known allergic sensitivity to EMLA cream® or amide type of local anaesthetics.
3. Patients with sensory peripheral neuropathy of both lower limbs.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analogue Score(VAS) | At the end of the treatment (day 1)
  At the end of the treatment i.e.Pain VAS will be assessed 60 mins after application of the study cream

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wee Aw, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- University Dermatology Clinic, National University Hospital, Singapore, Singapore, Singapore